CLINICAL TRIAL: NCT03415048
Title: Longitudinal Study of Children With Concussions: 3-year Follow-up of Cognitive and Emotional Function, Return to Sports, and Risk of Re-injury
Brief Title: Longitudinal Study of Children With Concussions
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Cynthia LaBella, Attending Physician, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: IRB2014-15813
Record Dates: First submitted 2016-01-26; First posted 2018-01-30 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Concussions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No Intervention

SUMMARY:
For children and adolescents who have had a concussion resulting in prolonged symptoms (>3 months), the investigators will:

1. Measure post-concussion symptoms, cognitive and emotional function during the 3 years post-injury.
2. Determine length of recovery and frequency of return to prior level of sports participation.
3. Determine the incidence of and risk factors for subsequent concussion during the 3 years post-injury.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 8-17 years old who present to one of the Lurie Sports Medicine clinics for care of a concussion.
2. English-speaking patients

Exclusion Criteria:

1. Patients outside of the 8-17 years old age range
2. Patients who show structural abnormalities on neuroimaging.
3. Non-English speaking patients

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children Ages 8-17 who present to one of the Lurie Sports Medicine clinics for care of a concussion.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Long-Term Effects of Concussion | 3 years
  All of the following measures will be aggregated using PROMIS - a computerized survey tool: what sports are played by the participant, whether or not the participant has quit a sport (due to concussion or not), development of anxiety or depression post-concussion, changes in peer relations post-concussion, change in cognitive function post-concussion, and if the participant has been subjected to a stigma after being diagnosed with a concussion.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia LaBella, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States